CLINICAL TRIAL: NCT00002025
Title: Open Label Ganciclovir Therapy for Sight- or Life-Threatening Cytomegalovirus Disease in the Immunocompromised Patient
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: None | Purpose: Treatment
Other Study IDs: 029D; ICM 1691
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1989-09

CONDITIONS: Cytomegalovirus Infections; Cytomegalovirus Retinitis; HIV Infections
Keywords: Retinitis; AIDS-Related Opportunistic Infections; Immune Tolerance; Injections, Intravenous; Ganciclovir; Cytomegalovirus Infections; Acquired Immunodeficiency Syndrome
MeSH Terms: conditions — Cytomegalovirus Infections; Cytomegalovirus Retinitis; HIV Infections; Retinitis; AIDS-Related Opportunistic Infections; Multiple Acyl Coenzyme A Dehydrogenase Deficiency; Acquired Immunodeficiency Syndrome | interventions — Ganciclovir

INTERVENTIONS:
Drug: Ganciclovir

SUMMARY:
To make intravenous (IV) ganciclovir available to immunocompromised patients with life-threatening or sight-threatening Cytomegalovirus (CMV) infection, where the symptoms of the disease are too severe to allow admission to a controlled clinical study of ganciclovir therapy. To determine the safety and tolerance of 2 - 3 weeks induction course of ganciclovir IV followed by a maintenance course of ganciclovir IV for an indefinite duration. To tabulate the patient's clinical response.

ELIGIBILITY:
Exclusion Criteria

Co-existing Condition:

Patients with the following are excluded:

* Cytomegalovirus (CMV) disease who meet the criteria for a treatment IND protocol, or other clinical studies, including controlled clinical studies of anticytomegalovirus therapy in peripheral CMV retinitis in patients with AIDS.
* Mild to moderate CMV infections who fail to meet the severity criteria. CMV syndrome (i.e., cytopenia, increased liver enzymes, fever, viremia, viruria) is not considered immediately life-threatening.
* Transplant patients in whom trial reduction of immunosuppressive drug treatment is feasible.
* Children with congenital or neonatal CMV where there is not a documented primary or acquired immunodeficiency.
* Hypersensitivity to acyclovir or ganciclovir.
* Receiving antimetabolite treatment that cannot be discontinued.

Concurrent Medication:

Excluded:

* Antimetabolites.
* Alkylating agents.
* Nucleoside analogs (topical ophthalmics are permitted).
* Interferon.
* Foscarnet.
* Cytokines.

Patients with the following are excluded:

* Cytomegalovirus (CMV) infection who meet the criteria for a treatment IND protocol, or other clinical studies, including controlled clinical studies of anticytomegalovirus therapy in peripheral CMV retinitis in patients with AIDS.
* Mild to moderate CMV infections who fail to meet the severity criteria. CMV syndrome (i.e., cytopenia, increased liver enzymes, fever, viremia, viruria) is not considered immediately life-threatening.
* Transplant patients in whom trial reduction of immunosuppressive drug treatment is feasible.
* Children with congenital or neonatal CMV where there is not a documented primary or acquired immunodeficiency.
* Hypersensitivity to acyclovir or ganciclovir.
* Receiving antimetabolite treatment that cannot be discontinued.

Patients must qualify as follows:

* Previously enrolled in compassionate use study (ICM 1257/1257A) or have terminated from another Syntex ganciclovir study.
* Diagnosis of AIDS and life-threatening Cytomegalovirus (CMV) infection.
* Diagnosis of other immunodeficiencies other than AIDS, with life-threatening or sight-threatening CMV disease.

Min Age: 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Roche Global Development - Palo Alto, Palo Alto, California, United States